CLINICAL TRIAL: NCT04861389
Title: The Comparison of Distal Transradial Access and Transradial Access for Primary Percutaneous Coronary Intervention in STEMI Patients（RESERVE Trial） A Single-center, Open, Prospective, Randomized Controlled Trial
Brief Title: Distal Transradial Access for Primary Percutaneous Coronary Intervention in STEMI Patients
Acronym: RESERVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RESERVE.01
Record Dates: First submitted 2020-11-29; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction; Radial Artery Occlusion; Distal Radial Artery Approach
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Arterial Occlusive Diseases | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal transradial access (dTRA) (Experimental): Distal transradial access for primary percutaneous coronary intervention in STEMI patients
  Interventions: Procedure: Arterial access
- Transradial access (TRA) (Active Comparator): Transradial access for primary percutaneous coronary intervention in STEMI patients
  Interventions: Procedure: Arterial access

INTERVENTIONS:
Procedure: Arterial access — Arterial access for primary percutaneous coronary intervention in STEMI patients

SUMMARY:
The transradial access (TRA) is currently the preferred approach for percutaneous coronary intervention (PCI). However, in patients with ACUTE ST-segment elevation myocardial infarction (STEMI) after emergency PCI, the high incidence of THE radial artery RAO limits the future choice of the radial artery for percutaneous intervention. The literature reported that distal transradial access (dTRA) significantly reduced RAO after elective PCI, but the application of dTRA in emergency PCI in STEMI has not been reported. We have completed 126 cases of dTRA undergoing emergency PCI after STEMI, which has been preliminarily confirmed to be safe and effective. A single-center, open, prospective, randomized controlled study is planned to compare the use of dTRA and TRA in emergency PCI in STEMI patients. The primary endpoint was the INCIDENCE of RAO within 24 hours after surgery. This clinical study verified that dTRA compared with TRA could reduce the RAO incidence of STEMI patients after emergency PCI. The project will explore a new artery approach to reduce RAO, and provide a basis for the selection of artery approach in STEMI emergency PCI patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of STEMI
* To undergo emergency PCI treatment
* Palpable pulsation of the radial artery and distal radial artery

Exclusion Criteria:

* Arteriovenous fistula of radial artery and cephalic vein has been performed with regular hemodialysis
* Suspicious left main block of electrocardiogram
* Had used the radial artery percutaneous interventional treatment before
* Cardiogenic shock

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The RAO incidence during hospitalization | 7 days
  The incidence of radial artery occlusion during hospitalization

SECONDARY OUTCOMES:
Puncture time | During the intervention
  Puncture time
Compression time | 4-24 hours
  Compression time
Puncture success rate | During the intervention
  Puncture success rate
Incidence of hematoma, finger numbness or pain during hospitalization | 7days
  Incidence of hematoma, finger numbness or pain during hospitalization
Incidence of RAO at 1 and 6 months after surgery | 1 and 6 months
  Incidence of RAO at 1 and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shaohong Dong, MD, Study Chair — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No